CLINICAL TRIAL: NCT03070236
Title: PORTAL: Patient-reported Outcomes After Routine Treatment of Atypical Lesions
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Ann H. Partridge, MD, MPH, Director, Adult Survivorship Program, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-571
Record Dates: First submitted 2017-02-16; First posted 2017-03-03 (Actual); Results first posted 2020-03-09 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient-reported Outcomes Survey (Experimental): The survey will administered online, over the phone, or via mail.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Select questions will be ask in the survey

SUMMARY:
This research study is evaluating how patients feel physically and emotionally after a prior breast biopsy for specific breast conditions (including atypical lesions such as atypical ductal hyperplasia (ADH), atypical lobular hyperplasia (ALH), lobular carcinoma in situ (LCIS), and/or ductal carcinoma in situ (DCIS))

DETAILED DESCRIPTION:
The goal of this research is to better understand the experience of women who have been diagnosed with certain breast conditions to enable women (and their doctors) to make informed decisions about their care.

ELIGIBILITY:
Inclusion Criteria:

Patients treated at DUMC, DFCI, MDACC, MGH, NWH, or DFCI @ SSH with a diagnosis of DCIS, LCIS, ADH, or ALH who are also:

* Age 18 or more at index diagnosis
* Diagnosed with DCIS, LCIS, ADH, or ALH between January 1, 2012 and June 30, 2017
* Able to read either English or Spanish and able to provide written (via paper), or on-line informed consent
* Treated and followed at one of the study sites (including affiliated network sites) and for whom treatment and surveillance data are available, for at least 1 year of follow up after date of diagnosis
* Participants with bilateral synchronous or metachronous disease (DCIS, LCIS, ADH, ALH) are eligible

Exclusion Criteria:

* Ever had a diagnosis of invasive or microinvasive breast cancer
* DCIS prior to index lesion or history of progressive/recurrent DCIS after treatment
* Other cancers (excluding non-melanoma skin cancer) diagnosed within 5 years prior to index lesion, including concurrent invasive cancer diagnosis and up to the present time of participant's approach to invitation into the study
* Patients identified by treating physician as being unsuitable for contact

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 912 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-05-27 (Actual); Study Completion 2030-02-25 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ann H. Partridge, MD, MPH, Study Director — Dana-Farber Cancer Institute
Locations (6):
- United States (6):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center in clinical affiliation with South Shore Hospital, Weymouth, Massachusetts
  - Duke University Medical Center, Durham, North Carolina
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Guideline Concordant Care (GCC) & Active Surveillance (AS): Guideline Concordant Care (GCC): Women who receive a combination of surgery, radiation and hormonal therapy - treatments similar to those recommended to patients with invasive cancer.
  Active Surveillance (AS): Women who receive a treatment strategy, under study for management of low-risk DCIS, that does not include surgery or radiation.
Period: Overall Study
Arm/Group | Guideline Concordant Care (GCC) & Active Surveillance (AS)
Started | 912
Guideline Concordant Care (GCC) arm | 538
Active Surveillance (AS) arm | 374
Completed | 912
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Guideline Concordant Care (GCC): Women who receive a combination of surgery, radiation and hormonal therapy - treatments similar to those recommended to patients with invasive cancer.
- Active Surveillance (AS): Women who receive a treatment strategy, under study for management of low-risk DCIS, that does not include surgery or radiation.
- Total: Total of all reporting groups
Arm/Group | Guideline Concordant Care (GCC) | Active Surveillance (AS) | Total
Number analyzed (Participants) | 538 | 374 | 912
Age, Continuous [Mean (Full Range); unit: years] | 60.7 [34.4 to 88.2] | 58.4 [26.1 to 94.1] | 59.8 [26.1 to 94.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 538 | 374 | 912
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 19 | 50
  Not Hispanic or Latino | 503 | 350 | 853
  Unknown or Not Reported | 4 | 5 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 22 | 20 | 42
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 40 | 15 | 55
  White | 459 | 330 | 789
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 17 | 9 | 26
Region of Enrollment [Number; unit: participants]
  United States | 538 | 374 | 912

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Measures Severity of Chronic Pain.
Description: The Breast Cancer Pain Questionnaire (BCPQ) is a validated, self-reported instrument assessing pain severity, pain frequency (how many days per week), and pain location (breast, arm, side, axilla) over the last 2-week period with an average of 45.8 months from treatment for the two groups, Guideline Concordant Care (GCC) and Active Surveillance (AS). The Pain Burden Index (PBI) is a composite of pain severity, pain frequency, and pain location. Each severity answer is multiplied by each frequency answer and then summed with a total possible score ranging from 0-200 with higher scores indicating worse pain.
Time Frame: Patient reported outcome was scheduled from at least one year from diagnosis. Participants' time from diagnosis to completing a survey was an average of 45.8 months in this study cohort.
Measure: Mean (Full Range); unit: Composite Score
Arm/Group | Guideline Concordant Care (GCC) | Active Surveillance (AS)
Number analyzed (Participants) | 538 | 374
Composite Score | 6.4 [0.0 to 80.0] | 3.0 [0.0 to 64.0]

ADVERSE EVENTS:
Time Frame: Approximately 19 months
Arm/Group | Guideline Concordant Care (GCC) & Active Surveillance (AS)
All-Cause Mortality (participants affected / at risk) | 0/912
Serious Adverse Events (participants affected / at risk) | 0/912
Other Adverse Events (participants affected / at risk) | 0/912

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-05-20): https://cdn.clinicaltrials.gov/large-docs/36/NCT03070236/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-20): https://cdn.clinicaltrials.gov/large-docs/36/NCT03070236/SAP_001.pdf